CLINICAL TRIAL: NCT02802475
Title: Antibodies Causing Epilepsy Syndromes: The ACES Study.
Acronym: ACES
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Nationaal Epilepsie Fonds (Unknown)
Responsible Party: Principal Investigator, M.J. Titulaer, MD. PhD., Erasmus Medical Center
Other Study IDs: MEC 2014-463
Record Dates: First submitted 2016-06-07; First posted 2016-06-16 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Auto-immune Encephalitis; Epilepsy
Keywords: antibodies; auto-immune encephalitis; epilepsy; limbic encephalitis
MeSH Terms: conditions — Epilepsy; Limbic Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and (if available) CSF

GROUPS / COHORTS (2):
- acquired chronic, focal, epilepsy: patients ≥18 years of age, with acquired chronic epilepsy of unknown origin
  Interventions: Biological: vena punction
- new onset epilepsy: patients ≥18 years of age, with new onset status epilepticus or new onset seizures with suspicion of limbic encephalitis
  Interventions: Biological: vena punction

INTERVENTIONS:
Biological: vena punction

SUMMARY:
The Antibodies Causing Epilepsy Syndromes (ACES) Study is a observational cohort study focusing on detection of auto-immune epilepsy in patients with epilepsy of unknown origin.

DETAILED DESCRIPTION:
Recently new treatable causes of epilepsy have been identified. These disorders are caused by a disruption of the balance in the brain caused by inflammation. This inflammatory reaction is caused by an autologous reaction of the immune system to specific brain proteins. The body produces antibodies to specific parts of the brain. These disorders can lead to epilepsy, memory dysfunction and psychiatric problems. Recognition is necessary for good treatment. Mostly anti-epileptic drugs are insufficient. These diseases can be treated with immune-modulating therapy. The ACES Study will focus on determining the frequencies of known antibodies and finding new, currently unknown, antibodies, causing epilepsy. Therefore patients will be investigated with epilepsy of unknown origin. To find new antibodies sera of patients with epilepsy will be added to brain sections of rats and to cultivated neuronal cells to look for a reaction. If new antibodies will be detected clinical features will be mapped of the patients. Also effects of antibodies on brain cells will be determined. Discovery of new antibodies can provide new treatment options for these patients. Also it will enable to discover more about the pathologic mechanisms of epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 and older.
* Status epilepticus or new onset seizures with signs of limbic encephalitis (clinical picture, MRI (FLAIR abnormalities), EEG abnormalities or CSF findings (CSF pleocytosis, increased IgG index, oligoclonal bands), or:
* Patients with acquired chronic focal epilepsy with an unknown cause.

Exclusion Criteria:

* Children
* Epilepsy with known cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with acquired chronic focal epilepsy without known cause or new onset status epilepticus or new onset seizures with signs of encephalitis and unknown cause.
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
frequency of patients with known and novel antibodies | 3 year
  detection of specific known and novel, currently unknown, auto-antibodies by immunohistochemistry, live hippocampal neuron cultures and cell-based assay

SECONDARY OUTCOMES:
modified Rankin scale | 1 year
  outcome 1 year after inclusion in the study
Seizure frequency | 1 year
  seizure frequency 1 year after inclusion in the study
Treatment response | 3 months
  frequency of objective improvement of outcome (seizure frequency, modified Rankin Scale) after immunotherapy, as compared to matched controls (without antibodies) from our study to exclude an effect due to regression to the mean or natural nistory.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten J Titulaer, MD,PhD, Principal Investigator — Erasmus Medical Center
Locations (8):
- Netherlands (8):
  - Epilepsiecentrum Kempenhaeghe, Heemstede
  - Stichting Epilepsie Instelling Nederland (SEIN), Heemstede
  - Academic Hospital Maastricht, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Haga Hospital, The Hague
  - St. Elisabeth Hospital, Tilburg
  - UMCU, Utrecht